CLINICAL TRIAL: NCT03974633
Title: A Randomized Controlled Trial Evaluating Three Non-invasive Analgesic Techniques in Pain Prevention During Injections
Brief Title: Evaluation of Three Non-invasive Analgesic Techniques in Pain Prevention During Injections
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Enrique Salmeron (Other)
Responsible Party: Sponsor-Investigator, Enrique Salmeron, Principal Investigator, Instituto de Investigacion Sanitaria La Fe
Organization: Instituto de Investigacion Sanitaria La Fe (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2018/0547
Record Dates: First submitted 2019-05-28; First posted 2019-06-05 (Actual); Last update posted 2019-08-22 (Actual); Status verified 2019-08

CONDITIONS: Injection Pain Prevention
Keywords: Analgesia; Cryoanalgesia; Vibration analgesia; Local anesthetic
MeSH Terms: conditions — Agnosia | interventions — Injections

STUDY DESIGN:
Intervention Model Description: All subjects received four injections of 0,1mL of physiologic saline (0,9%NaCl) in the forehead, 2cm above the eyebrows, with a 29G needle, after applying each one of the 4 non-invasive anesthetic methods studied in the trial, except for the control zone. The anesthetic method utilized in each part of the forehead of each patient was randomized through simple randomization.
Who Masked: Outcomes Assessor
Masking Description: Outcomes were studied by an investigator that did not participate in the practical part of the trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control (Placebo Comparator): A subcutaneous injection of 0,1mL saline (0,9%NaCl) was administered in a part of the forehead, without administering any type of non-invasive analgesic
  Interventions: Combination Product: Injection
- Vibration (Experimental): A subcutaneous injection of 0,1mL saline (0,9%NaCl) was administered in a part of the forehead, while applicating a vibrating device on the skin below the injection site, before and during injection.
  Interventions: Combination Product: Injection
- Cold (Experimental): A subcutaneous injection of 0,1mL saline (0,9%NaCl) was administered in a part of the forehead, after applicating a bag of 50mL of frozen physiologic saline covered with a plastic glove on the injection site for 50 seconds
  Interventions: Combination Product: Injection
- Anesthetic cream (Experimental): subcutaneous injection of 0,1mL saline (0,9%NaCl) was administered in a part of the forehead, after applicating a uniform thickness of 2mm of the anesthetic cream EMLA covered with an adhesive transparent plastic dressing for 30 minutes
  Interventions: Combination Product: Injection

INTERVENTIONS:
Combination Product: Injection — All information is included in the Arm/group descriptions

SUMMARY:
Injections are associated to a certain level of pain which tolerance can vary between individuals. As regards non-invasive pain control techniques in subcutaneous injections, scarce literature exists with adequate levels of evidence and design quality to support any specific analgesic method.

In this study, the investigators evaluated the effectivity of three non-invasive analgesic techniques (cold, anesthetic cream and vibration) when performing subcutaneous forehead injections, in a series of 100 healthy volunteers.

DETAILED DESCRIPTION:
This study is a randomized, controlled, simple-blind clinical trial, and it has been approved by the Ethics Committee of the Medical Research Institute Hospital La Fe. The study included 100 healthy volunteered, and it was performed in the University and Polytechnic Hospital La Fe, Valencia.

The procedures of the study consisted in the sequential performance of four injections of 0,1mL of physiologic saline (0,9%NaCl) in the forehead of each subject, 2cm above the eyebrows, with a 29G needle, after applying any of the non-invasive anesthetic methods studied in the trial, except for the control zone. The anesthetic method utilized in each part of the forehead of each patient was randomized through simple randomization. Injections always started from the right side of the forehead to the left. The non-invasive analgesic methods utilized were:

* Control zone: None
* Vibration: Application of the vibrating device on the skin below the injection site, before and during injection.
* Cold: Application of a bag of 50mL of frozen physiologic saline covered with a plastic glove on the injection site for 50 seconds prior to performing the injection.
* Anesthetic cream: Application of a uniform thickness of 2mm of the anesthetic cream EMLA covered with an adhesive transparent plastic dressing for 30 minutes, before injection.

ELIGIBILITY:
Inclusion Criteria:

* Every subject who did not meet any of the exclusion criteria, and signed the informed consent, was included in the study

Exclusion Criteria:

* Subjects younger than 18
* Subjects that suffered from any local or systemic sensitivity alteration
* Subjects that suffered from any cognitive deficit
* Individuals allergic to any of the components of the anesthetic ointment EMLA (eutectic mixture of lidocaine 2,5% and prilocaine 2,5%).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2018-02-24 (Actual); Primary Completion 2019-04-22 (Actual); Study Completion 2019-05-01 (Actual)

PRIMARY OUTCOMES:
Pain referred per each zone injected: VAS | 1 hour max
  Pain measured through a Visual Analogic Scale with values from 0 to 10; being 0 complete absence of pain, and 10 the worst pain ever experienced.

SECONDARY OUTCOMES:
Discomfort associated to non-invasive analgesic techniques | 1 hour max
  Discomfort associated to non-invasive analgesic techniques. Direct question in the survey in which answer options were each one of the non-invasive analgesic techniques (Cold, VIbration, Anesthetic cream)
Preference of non-invasive analgesic technique | 1 hour max
  Preference of non-invasive analgesic technique. Direct question in the survey in which possible answer options were each one of the non-invasive analgesic techniques (Cold, VIbration, Anesthetic cream)

CONTACTS AND LOCATIONS:
Overall Officials: Enrique Salmeron-Gonzalez, MD, Principal Investigator — University and Polytechnic Hospital La Fe
Locations (1):
- University and Polytechnic Hospital La Fe, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Babamiri K, Nassab R. The evidence for reducing the pain of administration of local anesthesia and cosmetic injectables. J Cosmet Dermatol. 2010 Sep;9(3):242-5. doi: 10.1111/j.1473-2165.2010.00503.x. PMID 20883298
- [Background] Davoudi A, Rismanchian M, Akhavan A, Nosouhian S, Bajoghli F, Haghighat A, Arbabzadeh F, Samimi P, Fiez A, Shadmehr E, Tabari K, Jahadi S. A brief review on the efficacy of different possible and nonpharmacological techniques in eliminating discomfort of local anesthesia injection during dental procedures. Anesth Essays Res. 2016 Jan-Apr;10(1):13-6. doi: 10.4103/0259-1162.167846. PMID 26957683
- [Background] Strazar AR, Leynes PG, Lalonde DH. Minimizing the pain of local anesthesia injection. Plast Reconstr Surg. 2013 Sep;132(3):675-684. doi: 10.1097/PRS.0b013e31829ad1e2. PMID 23985640
- [Background] Taddio A, Lord A, Hogan ME, Kikuta A, Yiu A, Darra E, Bruinse B, Keogh T, Stephens D. A randomized controlled trial of analgesia during vaccination in adults. Vaccine. 2010 Jul 19;28(32):5365-9. doi: 10.1016/j.vaccine.2010.05.015. Epub 2010 May 16. PMID 20483194
- [Background] Ernst E, Fialka V. Ice freezes pain? A review of the clinical effectiveness of analgesic cold therapy. J Pain Symptom Manage. 1994 Jan;9(1):56-9. doi: 10.1016/0885-3924(94)90150-3. PMID 8169463
- [Background] Elibol O, Ozkan B, Hekimhan PK, Caglar Y. Efficacy of skin cooling and EMLA cream application for pain relief of periocular botulinum toxin injection. Ophthalmic Plast Reconstr Surg. 2007 Mar-Apr;23(2):130-3. doi: 10.1097/IOP.0b013e318030459c. PMID 17413628
- [Background] Simons FE, Gillespie CA, Simons KJ. Local anaesthetic creams and intradermal skin tests. Lancet. 1992 May 30;339(8805):1351-2. doi: 10.1016/0140-6736(92)91994-j. No abstract available. PMID 1350007
- Available data/document: Individual Participant Data Set — https://docs.google.com/spreadsheets/d/1dEjSUmhIkqAOvh30WaJ0svs6jrdEGDyU5FXHeBuTOF8/edit?usp=sharing

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-19): https://cdn.clinicaltrials.gov/large-docs/33/NCT03974633/Prot_SAP_001.pdf